CLINICAL TRIAL: NCT01253759
Title: 10 Years Report of Combined Simultaneous Transpupillary Thermotherapy and ICG-based Photodynamic Therapy for Choroidal Melanoma
Brief Title: Long Term Results of Combined Transpupillary Thermotherapy (TTT) Indocyanine Green (ICG) Based Photodynamic Therapy (PDT) in Choroidal Melanoma
Status: Completed | Type: Observational
Sponsor: New England Retina Associates (Other)
Responsible Party: Principal Investigator, Peter E. Liggett, Principal Investigator, New England Retina Associates
Other Study IDs: NERA-2
Record Dates: First submitted 2009-03-25; First posted 2010-12-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Choroidal Melanoma
Keywords: Transpupillary thermotherapy; Choroidal melanoma; ICG-Photodynamic therapy
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Combined treatment of Transpupillary Thermotherapy and ICG-based photodynamic therapy (PDT)
  Interventions: Procedure: TTT + ICG-based PDT

INTERVENTIONS:
Procedure: TTT + ICG-based PDT

SUMMARY:
This is a report of 10 years results of combined Transpupillary thermotherapy (TTT) treatment with Indocyanine green (ICG) in controlling small and medium-sized choroidal melanomas.

DETAILED DESCRIPTION:
The study was done in a Clinical practice setting. Forty six eyes of 46 patients with small or medium-sized choroidal melanomas were treated with i-TTT using infrared light delivered from a diode laser. All patients were evaluated to rule out systemic metastasis and underwent a complete ophthalmological evaluation including: Slit lamp biomicroscopy, dilated fundus examination, Fluorescein angiography, Optical coherence tomography and A/B ultrasonography. Main outcome measures were: Changes in visual acuity, complications associated with the treatment and local control of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Small and medium-sized choroidal melanoma
* Patients older than 18 years old.
* Patients who can read and signed the informed consent.

Exclusion Criteria:

* Patients with ocular inflammation.
* Patients with another active ocular disease.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects selected from retina specialist general patient population.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter E Liggett, MD, Study Director — New England Retina Associates
Locations (1):
- New England Retina Associates, Hamden, Connecticut, United States